CLINICAL TRIAL: NCT01025830
Title: Steady State Bioequivalence of Generic and Innovator Formulations of Stavudine, Lamivudine, and Nevirapine in HIV-infected Ugandan Adults
Brief Title: Triomune Bioequivalence With Innovators
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Jayne Tusiime, University of California, Berkeley
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BETr
Record Dates: First submitted 2009-04-21; First posted 2009-12-04 (Estimated); Results first posted 2009-12-04 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-12

CONDITIONS: HIV/AIDS
Keywords: HIV;Bioequivalence;Triomune
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — stavudine, lamivudine, nevirapine drug combination; Stavudine; Lamivudine; Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic (Experimental): generic fixed dose combination of Stavudine, Lamivudine and Nevirapine (Triomune)
  Interventions: Drug: Triomune
- Brand (Active Comparator): 3 separate single pills of Zerit (Stavudine)Epivir (Lamivudine) Viramune (Nevirapine)
  Interventions: Drug: Zerit/Epivir/Viramune

INTERVENTIONS:
Drug: Triomune — Stavudine (40mg) Lamivudine (150mg) Nevirapine (200mg)All twice a day
  Other Names: Stavudine; Lamivudine; Nevirapine
  Arms: Generic
Drug: Zerit/Epivir/Viramune — Stavudine (40mg) Lamivudine (150mg) and Nevirapine (200mg) All taken twice daily.
  Other Names: Stavudine; Lamivudine; Nevirapine
  Arms: Brand

SUMMARY:
The null hypothesis is that there is a difference in the the relative rate and extent of absorption into the systemic circulation of Triomune and brand-name Stavudine/Lamivudine/Nevirapine in HIV-infected Africans and the alternative hypothesis is that there is no difference in the the relative rate and extent of absorption into the systemic circulation of Triomune and brand-name Stavudine/Lamivudine/Nevirapine in HIV-infected Africans. This is a non-inferiority study.

DETAILED DESCRIPTION:
Generic antiretroviral therapy is the mainstay of HIV treatment in resource-limited settings, yet there is little evidence confirming the bioequivalence of generic and brand name formulations. We compared the steady-state pharmacokinetics of Lamivudine, Stavudine and Nevirapine in HIV-infected subjects who were receiving a generic formulation (Triomune®) or the corresponding brand formulations (Epivir®, Zerit®, and Viramune®). An open-label, randomized, crossover study was carried out in 18 HIV-infected Ugandan subjects stabilized on Triomune-40. Subjects received Lamivudine (150 mg), Stavudine (40 mg), and Nevirapine (200 mg) in either the generic or brand formulation twice a day for 30 days, before switching to the other formulation. At the end of each treatment period, blood samples were collected over 12 h for pharmacokinetic analysis. The main outcome measures were the mean AUC0-12h and Cmax. Bioequivalence was defined as a geometric mean ratio between the generic and brand-name within the 90% confidence interval of 0.8-1.25.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected men and non-pregnant women;
2. On Triomune for at least 4 weeks;
3. 18 years or greater;
4. Residing within 15km of Kampala city center

Exclusion Criteria:

1. Unable to sign or understand informed consent
2. Concurrent medication known to interact with any of the components of Triomune
3. Patients with active TB, malabsorption, nausea, emesis, abdominal discomfort, chronic diarrhoea, documented active clinically relevant hepatitis;
4. Patients expected to change their drug regimen or dosage during the study
5. Those planning to move out of Kampala in the next two months;
6. Hemoglobin <7.0 mmol/l (men) or <6.5 mmol/l (women);
7. Alanine aminotransferase or aspartate aminotransferase >5 times the upper limit of normal;
8. Serum creatinine > 1.5 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02; Primary Completion 2006-06 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Tusiime, B Pharm, MSc, Principal Investigator — Makerere University; David R Bangsberg, MD,MPH, Study Chair — Harvard University
Locations (1):
- Makerere University, Kampala, Uganda

REFERENCES:
- [Result] Byakika-Tusiime J, Chinn LW, Oyugi JH, Obua C, Bangsberg DR, Kroetz DL. Steady state bioequivalence of generic and innovator formulations of stavudine, lamivudine, and nevirapine in HIV-infected Ugandan adults. PLoS One. 2008;3(12):e3981. doi: 10.1371/journal.pone.0003981. Epub 2008 Dec 19. PMID 19096711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from an ongoing cohort study in Kampala, Uganda. The first subject was recruited in Feb 2006.
Pre-assignment Details: Participants received a medical and laboratory examination before assignment. Subjects were excluded if they had active tuberculosis or were anemic. 22 participants were recruited; 22 were screened,2 were excluded (1 did not meet inclusion criteria and 1 refused participation).
Groups:
- Generic (Triomune) to Brand (Zerit/Epivir/Viramune): Started with generic formulation (Triomune) then switched to brand formulation (Zerit/Epivir/Viramune).
- Brand (Zerit/Epivir/Viramune) to Generic (Triomune): started with brand formulation(Zerit/Epivir/Viramune) then switched to generic formulation (Triomune)
Period: Generic (Tr) First Then Brand (Ze/Ep/Vi)
Arm/Group | Generic (Triomune) to Brand (Zerit/Epivir/Viramune) | Brand (Zerit/Epivir/Viramune) to Generic (Triomune)
Started | 8 | 12
Completed | 8 | 12
Not Completed | 0 | 0
Period: Washout Period of 30 Days
Arm/Group | Generic (Triomune) to Brand (Zerit/Epivir/Viramune) | Brand (Zerit/Epivir/Viramune) to Generic (Triomune)
Started | 8 | 12
Completed | 8 | 12
Not Completed | 0 | 0
Period: Brand (Ze/Ep/Vi) First Then Generic (Tr)
Arm/Group | Generic (Triomune) to Brand (Zerit/Epivir/Viramune) | Brand (Zerit/Epivir/Viramune) to Generic (Triomune)
Started | 8 | 12
Completed | 8 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive generic formulation and brand formulation
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.1 (3.4)
Weight [Mean (Standard Deviation); unit: kg] | 68.3 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve(AUC)
Description: Mean Area Under the Plasma Concentration-Time Curve for each drug, log transformed
Time Frame: Assessed at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 10 and 12 hr post-dosing
Population: Analyzed population consists only of participants who had sufficient plasma samples for analysis.Intent to treat analysis was used. Separate analyses provided for each drug. Results of such a study are not combined.
Measure: Geometric Mean (Standard Deviation); unit: hour*milligram/liter
Groups:
- Generic Stavudine: period when subjects were on generic stavudine
- Brand Stavudine: period when subjects were on brand stavudine
- Generic Nevirapine: period when subjects were on generic nevirapine
- Brand Nevirapine: Period when subjects were on brand nevirapine
- Generic Lamivudine: period when subjects were on generic lamivudine
- Brand Lamivudine: Period when subjects were on brand lamivudine
Arm/Group | Generic Stavudine | Brand Stavudine | Generic Nevirapine | Brand Nevirapine | Generic Lamivudine | Brand Lamivudine
Number analyzed (Participants) | 7 | 11 | 7 | 11 | 7 | 11
hour*milligram/liter | 3.6 (2.4) | 3.4 (3.9) | 85.8 (35.2) | 79.2 (45.7) | 5.2 (2.5) | 6.4 (4.9)
Statistical Analysis 1: Comparison: Generic Stavudine vs Brand Stavudine; The null hypothesis was that there is a difference in the relative bioavailability of Triomune and brand-name stavudine/lamivudine/nevirapine in HIV-infected Africans. 18 participants were required to provide 80% power to detect approximately a 20% difference on a log scale in AUC0-12h between the brand formulation and the generic formulation. Alpha level of 0.05; Test type: Non-Inferiority or Equivalence — Bioequivalence was defined as a 90% Confidence Interval of the geometric mean ratio between 0.8 and 1.25. Differences between treatments with respect to the outcome and intra- and inter-subject variances were assessed using the mixed effects model. Bootstrapped random errors were used; Non-compartmental model — p value not required for this analysis. What counts is the 90% confidence interval of the geometric mean ratio between the two formulation parameters; Mixed random effects model was used to assess difference between treatments and intra- and inter-subject variances; Geometric Mean Ratio = 1.1, 90% CI [0.87 to 1.38] — the generic is the numerator while the brand is the denominator
Statistical Analysis 2: Comparison: Generic Nevirapine vs Brand Nevirapine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Non-compartmental model — [p-value comment as in outcome 1, analysis 1]; Mixed random effects model was used to assess difference between treatments and intra- and inter-subject variances; Geometric Mean Ratio = 1.1, 90% CI [0.95 to 1.31] — the generic is the numerator while the brand is the denominator
Statistical Analysis 3: Comparison: Generic Lamivudine vs Brand Lamivudine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Non-compartmental model — [p-value comment as in outcome 1, analysis 1]; Mixed random effects model was used to assess difference between treatments and intra- and inter-subject variances; Geometric Mean Ratio = 0.8, 90% CI [0.65 to 0.99] — the generic is the numerator while the brand is the denominator

2. Secondary Outcome: Maximum Plasma Concentration of Drug
Description: Maximum concentration of drug in plasma that was attained post dosing
Time Frame: Assessed at 0, 0.5, 1, 1.5, 2, 3, 4, 6, 10 and 12 hr post-dosing
Population: Intention to treat analysis used including only participants with sufficient plasma samples for analysis. Separate analyses are given for each drug. Results for this kind of study are not combined.
Measure: Geometric Mean (Standard Deviation); unit: milligram/liter
Arm/Group | Generic Stavudine | Brand Stavudine | Generic Nevirapine | Brand Nevirapine | Generic Lamivudine | Brand Lamivudine
Number analyzed (Participants) | 7 | 11 | 7 | 11 | 7 | 11
milligram/liter | 1.6 (1.1) | 1.3 (2.0) | 8.8 (3.1) | 8.4 (5.5) | 1.0 (0.5) | 1.3 (1.4)
Statistical Analysis 1: Comparison: Generic Stavudine vs Brand Stavudine; Same as for AUC; Test type: Non-Inferiority or Equivalence — same as for AUC; Non-compartmental model — same as for AUC; same as for AUC; Geometric Mean Ratio = 1.3, 90% CI [0.99 to 1.71] — same as AUC
Statistical Analysis 2: Comparison: Generic Nevirapine vs Brand Nevirapine; Same for all three drugs; Test type: Non-Inferiority or Equivalence — same for all three drugs; Non-compartmental model — Same for all three drugs; Same for all three drugs; Geometric Mean Ratio = 1.1, 90% CI [0.95 to 1.23] — Same for all three drugs
Statistical Analysis 3: Comparison: Generic Lamivudine vs Brand Lamivudine; Same for all three drugs; Test type: Non-Inferiority or Equivalence — Same for all three drugs; Non-compartmental model — Same for all three drugs; Same for all three drugs; Geometric Mean Ratio = 0.8, 90% CI [0.63 to 0.98] — Same for all three drugs

ADVERSE EVENTS:
Time Frame: Patients were in the study for 60 days and this is the period over which they were monitored for any adverse events.
Description: After 30 days of taking each formulation subjects were asked if they had experienced any unwanted effects since they started taking the study drug. Responses were recorded in their study charts. During the blood draw period patients were watched for any adverse events.
Groups:
- Generic to Brand: Started with generic formulation then switched to brand formulation
- Brand to Generic: started with brand formulation then switched to generic formulation
Arm/Group | Entire Study Population | Generic to Brand | Brand to Generic
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 0/20 | 0/8 | 0/12

LIMITATIONS AND CAVEATS:
Stavudine (40mg) was used whereas currently it is Stavudine(30mg) that is recommended for usage. So our results may not be applicable to patients on Stavudine 30mg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No